CLINICAL TRIAL: NCT02498314
Title: Clinical Effects of Translatoric Grades of Movement in Hip Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Elena Estebanez de Miguel, Unidad de investigación en Fisioterapia, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI11/00061; PUZ/1 (Other: Universidad de Zaragoza)
Record Dates: First submitted 2015-07-08; First posted 2015-07-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Hip Osteoarthritis
Keywords: Manual therapy; Hip osteoarthritis; Mobilization
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Grade I-II SZ mobilization (Experimental): Grade I-IISZ hip traction in resting position
  Interventions: Other: Grade I-II SZ mobilization
- Grade II TZ mobilization (Experimental): Grade IITZ hip traction in resting position
  Interventions: Other: Grade II TZ mobilization
- Grade III mobilization (Experimental): Grade III hip traction in resting position
  Interventions: Other: Grade III mobilization

INTERVENTIONS:
Other: Grade I-II SZ mobilization — Hip grade I-IISZ traction in a resting position is applied using gentle repetitive traction movements during 10 minutes. The mean peak force applied is 2,71N (S.D= 0,94), according to previous study. Peak forces were measured using dynamometer and the therapist used it as a feedback to ensure mean peak force levels remain consistent.
  Arms: Grade I-II SZ mobilization
Other: Grade II TZ mobilization — Hip grade IITZ traction in a resting position is applied during 10 minutes. The traction force is applied during 45 seconds with 15 seconds rest, until complete the 10 minutes of treatment. The mean peak force applied is 5.94 N (S.D= 1), according to previous study. Peak forces were measured using dynamometer and the therapist used it as a feedback to ensure mean peak force levels remain consistent.
  Arms: Grade II TZ mobilization
Other: Grade III mobilization — Hip grade III traction in a resting position is applied during 10 minutes. The traction force is applied during 30 seconds with 30 seconds rest, until complete the 10 minutes of treatment. The mean peak force applied is 7.04 N (S.D= 0.32), according to previous study. Peak forces were measured using dynamometer and the therapist used it as a feedback to ensure mean peak force levels remain consistent.
  Arms: Grade III mobilization

SUMMARY:
In orthopaedic manual therapy translatoric grades of movement are used to determine the intensity of force applied during the mobilization. Different clinical effects are described for each translatoric grade of movement but there are not published studies evaluating these clinical effects.

The objective of this trial is to determine if force magnitude during hip traction in resting position affects immediate and short-term outcomes (pain, physical function, hip muscle length and hip range of motion) in patients with hip osteoarthritis. For this purpose, investigators conduct a randomized clinical trial, double-blind (patient and physical therapist examiner). Participants entering the study were randomized into 1 of 3 treatment groups: grade I- grade IISZ mobilization, grade IITZ mobilization or grade III mobilization. Participants attend three sessions on alternate days (monday, wednesday, friday) and at the same hour. Measurements are taken prior to treatment, immediately after each session treatment.

The participants are recruited from physiotherapy groups or referred by general practitioners and orthopedic surgeons.

Participants were assigned to 1 of the 3 study groups through concealed allocation (sealed envelopes) and independent blocked randomization, using a random number generator.

One physical therapist enroll patients in the study, while an independent research assistant performed the randomization and prepared the sealed envelopes, which are opened after baseline data collection by the physiotherapist performing the treatments. Participants are treated in a private treatment area and have no knowledge of treatments received by other participants.

A second experienced orthopaedic manual therapist applies the standardized hip traction mobilization in resting position at either level of force, during 10 minutes. This amount of mobilization is consistent with clinical practice and previous studies in osteoarthritis patients.

Two physiotherapists (third and fourth) with 5 years of experience, who were blinded to participant group, performed all measurements.The outcome measures are pain, physical function, hip muscle length and hip passive range of motion. Pain is registered with visual analogic scale (VAS), Pressure Pain Threshold ( PPT) and WOMAC pain subscale. Physical function is registered using Timed Up & Go test (TUG), the 20-Meter Walking Test (20MWT) and the physical function subscale of WOMAC index. The hip muscle length is measured using Ely´s test, Active Knee Extension test and modified Ober´s test. The passive hip range of motion is measured using inclinometer or goniometer.

ELIGIBILITY:
Inclusion Criteria:

* unilateral primary hip OA according to the clinical criteria of the American College of Reumathology,
* a grade III Kellgren & Lawrence (K-L) classification in their most recent hip X-rays,
* mild to moderate pain from hip OA categorized using the WOMAC pain subscale (2 to 8 as mild pain; greater than 8 to 12 as moderate pain),
* the ability to walk at least 20 meters, with or without an aid.

Exclusion Criteria:

* neurological, vascular or other lower extremity musculoskeletal conditions that affected sensation, gait or functional performance,
* contraindications for manual therapy
* insufficient understanding of the Spanish language

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain on the VAS scale | pre-intervention and post-intervention (baseline and 5 days)
Pressure Pain Threshold (PPT) | pre-intervention and post-intervention (baseline and 5 days)
Pain on the pain subscale of WOMAC index (WOMAC-P) | pre-intervention and the next day of the last treatment session (baseline and 6 days)

SECONDARY OUTCOMES:
Physical Function on Timed Up & Go test (TUG) | pre-intervention and post-intervention (baseline and 5 days)
Physical Function on the 20-Meter Walking Test | pre-intervention and post-intervention (baseline and 5 days)
Physical Function on The physical function subscale of WOMAC index (WOMAC-PF) | pre-intervention and the next day of the last treatment session (baseline and 6 days)
Hip range of motion with digital inclinometer | pre-intervention and post-intervention (baseline and 5 days)
  Passive hip range of motion in the three planes is measured before and after each treatment sessions with a digital inclinometer
Rectus femoris flexibility assessment: Ely´s test | pre-intervention and post-intervention (baseline and 5 days)
Hamstring flexibility assessment: Active Knee test | pre-intervention and post-intervention after each session (baseline and 5 days)
Iliotibial band tightness assessment: modified Ober´s test | pre-intervention and post-intervention (baseline and 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Estebanez, PhD, Principal Investigator — Unidad de Investigación en Fisioterapia. Zaragoza, Zaragoza, Spain
Locations (1):
- Elena Estebanez de Miguel, Zaragoza, Spain

REFERENCES:
- [Derived] Estebanez-de-Miguel E, Fortun-Agud M, Jimenez-Del-Barrio S, Caudevilla-Polo S, Bueno-Gracia E, Tricas-Moreno JM. Comparison of high, medium and low mobilization forces for increasing range of motion in patients with hip osteoarthritis: A randomized controlled trial. Musculoskelet Sci Pract. 2018 Aug;36:81-86. doi: 10.1016/j.msksp.2018.05.004. Epub 2018 May 29. PMID 29864710